CLINICAL TRIAL: NCT03788616
Title: Evaluation of Fluoride Release and Compressive Strength of a Bioactive Restorative Material and Its Clinical Performance in Atraumatic Restorative Treatment in Primary Molars (An in Vitro Study & A Randomized Controlled Trial )
Brief Title: Fluoride Release,Compressive Strength and Clinical Performance of a Bioactive Restorative Material in ART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marina F Fahmy, MD (Other)
Responsible Party: Sponsor-Investigator, Marina F Fahmy, MD, Assistant lecturer of pediatric dentistry, pediatric dentistry and public health department, Ain Shams University, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PED18-5M
Record Dates: First submitted 2018-12-14; First posted 2018-12-27 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries
Keywords: Bioactive Restorative Material , ART
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Group I : will consist of 30 teeth that will be restored by high-viscosity glass ionomer (Fuji IX Extra) with ART approach
  Interventions: Drug: Fuji IX EXTRA
- Group II (Active Comparator): Group II : will consist of 30 teeth that will be restored by bioactive restorative material (ACTIVA KIDS bioactive restorative material) with ART approach.
  Interventions: Drug: ACTIVA KIDS bioactive restorative material

INTERVENTIONS:
Drug: Fuji IX EXTRA — High-viscosity glass ionomer (Fuji IX EXTRA)
  Other Names: Extra fast GIC
  Arms: Group I
Drug: ACTIVA KIDS bioactive restorative material — Modified composite (ACTIVA KIDS)
  Other Names: ACTIVA , Modified composite
  Arms: Group II

SUMMARY:
The study will be two parallel group, triple blinded randomized controlled clinical trial that based on CONSORT (consolidated standards of reporting trials) guideline .The selected participants according to inclusion and exclusion criteria will be randomly allocated in two groups using (Research Randomizer Program) .

DETAILED DESCRIPTION:
Blinding All participants don't know the type of received restorative material (ACTIVA Kids or High -viscosity GI restorative material) and the outcome will be evaluated by a examiner other than operator who doesn't know the type of received restorative material also.

Study setting The study will be performed at pediatric Department and Dental Public Health Department of Faculty of Dentistry, Ain Shams University, and at the institute of Graduate Studies and Research, Ain Shams University.

Sample size: 60 participants Recruitment/Setting The all participants of this study have been selected after complete clinical examination has been done with full medical and dental history , history of medications and history of hospitalization. In patients who receive dental treatment as an usual care in clinics of Pediatric Dentistry and Dental Public Health Department at faculty of dentistry, Ain-Shams University.

Informed consent designed to include all data about dental procedures in this study and clear more details about time consuming in the procedure and follow up visits, used materials and adverse event of this procedure . All participants have the wright to withdraw from this study at any time .The consent will be assigned from each patient by the patient's parents or guardians after explanation of the study.

The full mouth rehabilitation will be performed by postgraduate student registered at the master Degree at the Pediatric Dentistry and Dental Public Health Department Faculty of Dentistry, Ain- Shams University All subjects receive instructions on oral health, particularly in relation to oral hygiene and sugar consumption

ELIGIBILITY:
Inclusion Criteria:

1. Children aged from 4 to 8 years old, in good general health
2. Children classified as class 3 or 4 based on Frankel et al. classification. (26)
3. The children have at least one primary molar with class I carious lesion.
4. Asymptomatic teeth (without spontaneous pain)

Exclusion Criteria:

1. Medically compromised patient
2. Presence of pulp exposure, pain, mobility
3. Presence of swelling, abscess or fistula near the tooth
4. Not accessible carious lesion to hand instruments

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2019-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amr Mahmoud Abd EL Aziz, Study Chair — Professor of Pediatric Dentistry and Dental Public Health Department -ASU; Reham Khaled Abou El Fadl, Study Director — Lecturer of Pediatric Dentistry and Dental Public Health Department -ASU
Locations (1):
- Marina Fakhry Fahmy Saad, Cairo, Egypt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients was done from a convenient sample of children who attended the outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Ain-Shams University seeking dental treatment, or for regular checkups. All patients who met the eligibility criteria of the study were invited to participate. Pre-operative comprehensive clinical examination was performed and caries experience was determined using dmft index
Pre-assignment Details: Excluded (n = 40)
  - Tooth not meeting inclusion criteria
Units Other Than Participants: primary molars
Groups:
- Fuji IX Extra Group I: Group I: will consist of 35 teeth that will be restored by high-viscosity glass ionomer (Fuji IX Extra) with an ART approach
  Fuji IX EXTRA: High-viscosity glass ionomer (Fuji IX EXTRA)
- Bioactive Composite Group II: Group II: will consist of 35 teeth that will be restored by bioactive restorative material (ACTIVA KIDS bioactive restorative material) with ART approach.
  ACTIVA KIDS bioactive restorative material: Modified composite (ACTIVA KIDS)
Period: Overall Study
Arm/Group | Fuji IX Extra Group I | Bioactive Composite Group II
Started | 35; 35 primary molars | 35; 35 primary molars
Completed | 30; 30 primary molars | 32; 32 primary molars
Not Completed | 5; 5 primary molars | 3; 3 primary molars

BASELINE CHARACTERISTICS:
Population: carious primary molars limited to occlusal table (class I cavity) in 4-8 yrs old patients
Units Other Than Participants: primary molars
Groups:
- Group I: Group I: will consist of 35 teeth that will be restored by high-viscosity glass ionomer (Fuji IX Extra) with ART approach
  Fuji IX EXTRA: High-viscosity glass ionomer (Fuji IX EXTRA)
- Group II: Group II: will consist of 35 teeth that will be restored by bioactive restorative material (ACTIVA KIDS bioactive restorative material) with ART approach.
  ACTIVA KIDS bioactive restorative material: Modified composite (ACTIVA KIDS)
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Total
Number analyzed (Participants) | 35 | 35 | 70
Number analyzed (primary molars) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: not meeting the inclusion criteria
  years | 5.6 (1.49) | 5.9 (1.49) | 5.7 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1. not meeting the inclusion criteria
  2. not complete the treatment plane
  Participants
    Female | 15 | 21 | 36
    Male | 20 | 14 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: the Success Rate of ACTIVA BIOACTIVE and Fuji IX Extra GIC With ART in Class I Carious Cavity of Primary Teeth
Description: Using Atraumatic restorative treatment criteria from 0 to 9, The restorations were considered to have survived when given scores 0,1, or 7 and to have failed with scores 2,3,4,8, while those scores 5,6 were considered to be unrelated to success and failure.
Time Frame: 12 Month
Measure: Number; unit: primary molars
Units Other Than Participants: primary molars
Groups:
- Fuji IX Extra GIC With ART: Group I: will consist of 35 teeth that will be restored by high-viscosity glass ionomer (Fuji IX Extra) with ART approach
  Fuji IX EXTRA: High-viscosity glass ionomer (Fuji IX EXTRA)
- ACTIVA KIDS With ART: Group II: will consist of 35 teeth that will be restored by bioactive restorative material (ACTIVA KIDS bioactive restorative material) with ART approach.
  ACTIVA KIDS bioactive restorative material: Modified composite (ACTIVA KIDS)
Arm/Group | Fuji IX Extra GIC With ART | ACTIVA KIDS With ART
Number analyzed (Participants) | 35 | 35
Number analyzed (primary molars) | 35 | 35
primary molars
  success rate after 3 Months | 30 | 32
  success rate after 6 months | 28 | 30
  success rate after 12 months | 26 | 25
Statistical Analysis 1: Comparison: Fuji IX Extra GIC With ART vs ACTIVA KIDS With ART; Test type: Equivalence — assuming 95% power of the study; p = 0.478, t-test, 2 sided; Median Difference (Final Values) = 0.05

ADVERSE EVENTS:
Time Frame: 3 months, 6 months,1 year
Description: failure of restorations in participated primary molars. (non-serious adverse event)
Groups:
- Fuji IX EXTRA GIC With ART: Group I : will consist of 35 teeth that will be restored by high-viscosity glass ionomer (Fuji IX Extra) with ART approach
  Fuji IX EXTRA: High-viscosity glass ionomer (Fuji IX EXTRA)
- ACTIVA KIDS With ART: Group II : will consist of 35 teeth that will be restored by bioactive restorative material (ACTIVA KIDS bioactive restorative material) with ART approach.
  ACTIVA KIDS bioactive restorative material: Modified composite (ACTIVA KIDS)
Arm/Group | Fuji IX EXTRA GIC With ART | ACTIVA KIDS With ART
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 4/35 | 7/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fuji IX EXTRA GIC With ART (N=35) | ACTIVA KIDS With ART (N=35)
failure of restoration (Product Issues) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03788616/Prot_SAP_000.pdf